CLINICAL TRIAL: NCT01833247
Title: Lactic Acidosis During and After Seizures
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert S. Fisher, M.D., Ph.D., Professor of Neurology, Stanford University
Other Study IDs: Stanford Epilepsy IRB 21989
Record Dates: First submitted 2013-03-28; First posted 2013-04-16 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
Keywords: epilepsy; lactic acid; saliva; postictal
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epilepsy inpatients: Patients with epilepsy recorded in an inpatient video-EEG monitoring unit after a seizure.

SUMMARY:
This project looks at the time course of lactic acid rise (if any) after seizures. Salivary and capillary lactic acid are tested. This type of measurement may be useful in signalling the occurrence or recent history of a seizure.

DETAILED DESCRIPTION:
Lactic acid is released from cells during seizures and elevates lactic acid levels in blood and saliva. The time course of this rise is unknown. If lactic acid rises within a few minutes of a seizure, than it might be feasible to develop lactic acid sensors to provide notification of a recent seizure. This could lead to better safety monitoring for people with epilepsy. This study was designed to utilize a commercially available lactic acid sensor (investigators have no connection with the sensor manufacturer and purchased the device at list price) to measure salivary lactic acid levels after a seizure during inpatient video-EEG epilepsy monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 inclusive.
2. History of at least one generalized tonic-clonic (grand mal) seizure prior to enrollment in the study.
3. Undergoing monitoring in the Stanford Epilepsy Monitoring Unit.

   Exclusion Criteria:
4. Not pregnant.
5. Inability to understand and sign the consent form.
6. No known history of mitochondrial disease or other metabolic disorders expected to affect blood lactate.
7. No known history of thrombophlebitis or excessive tendency to bleeding. Not on coumadin. Aspirin or anti-platelet agents are not an exclusion.
8. No known peripheral vascular disease affecting blood circulation to the fingers.
9. No painful peripheral neuropathy.
10. No Raynaud's disease or phenomenon.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age range will be 18-75, men and women, all ethnic backgrounds to be eligible. Eligible population will be determined by who gets admitted to the epilepsy monitoring unit with a history of generalized tonic-clonic seizures.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fisher, MD, PhD, Principal Investigator — Stanford University Department of Neurology
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
If subjects wish to know their lactic acid levels after a seizure, we will provide the information, although it currently has no therapeutic or prognostic implications.

RESULTS

PARTICIPANT FLOW:
Groups:
- Epilepsy Inpatients: Patients who have blood or salivary (or both) levels recorded after a seizure.
Period: Overall Study
Arm/Group | Epilepsy Inpatients
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with epilepsy in hospital for video-EEG recording
Arm/Group | Epilepsy Inpatients
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 40.8 [26 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Salivary Lactic Acid Levels With Seizures
Description: The investigators will assess the salivary lactic acid within 10 minutes after end of a seizure. Values will consist of lactic acid measurements in saliva , immediately post-seizure. Units of measurement will be mM/L. A positive outcome will be a curve different from a straight line, with a rise and fall of lactate levels. Baseline lactate serum level is expected to be less than 2.2 mM/L.
Time Frame: Within 10 minutes of end of the seizure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Epilepsy Inpatients
Number analyzed (Participants) | 12
mmol/L | 8.16 (8.88)

2. Primary Outcome: Capillary Lactic Acid Levels With Seizures
Description: The investigators will assess the capillary lactic acid within 10 minutes after end of a seizure. Values will consist of lactic acid measurements in blood, within 10 minutes after the end of a seizure. Units of measurement will be mM/L. Baseline lactate serum level is expected to be less than 2.2 mM/L.
Time Frame: Within 10 minutes of end of the seizure
Population: Data were collected from 6 of the 12 enrolled subjects
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Epilepsy Inpatients
Number analyzed (Participants) | 6
mmol/L | 5.67 (4.57)

3. Primary Outcome: Intravenous Lactic Acid Levels With Seizures
Description: The investigators will assess the intravenous lactic acid within 10 minutes after end of a seizure. Values will consist of lactic acid measurements in serum collected by IV, immediately post-seizure. Units of measurement will be mM/L. A positive outcome will be a curve different from a straight line, with a rise and fall of lactate levels. Baseline lactate serum level is expected to be less than 2.2 mM/L.
Time Frame: Within 10 minutes of end of the seizure
Population: Data were collected from one participant
Measure: Number; unit: mmol/L
Arm/Group | Epilepsy Inpatients
Number analyzed (Participants) | 1
mmol/L | 8.6

4. Post Hoc Outcome: Salivary and Capillary Lactic Acid Will be Correlated After a Seizure
Description: Salivary levels of lactic acid is being studied because saliva is more accessible in the outpatient setting than is blood. Concentration of lactic acid in the serum and saliva from each individual subject will be correlated using Pearson's correlation test. We will consider a positive outcome to be a r greater than or equal to 0.5 and significance at p<0.05.
Time Frame: Within 10 minutes of a seizure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Within 2 hours after the seizure
Arm/Group | Epilepsy Inpatients
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Salivary lactic acid levels were difficult to reliably obtain with commercial devices designed to measure blood salivary levels. Because of low reliability, we did not pursue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No